CLINICAL TRIAL: NCT01120470
Title: A Randomized Phase II Study of OGX-427 (a Second-Generation Antisense Oligonucleotide to Heat Shock Protein-27) in Patients With Castration Resistant Prostate Cancer Who Have Not Previously Received Chemotherapy for Metastatic Disease
Brief Title: OGX-427 in Castration Resistant Prostate Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: Achieve Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR-01
Record Dates: First submitted 2010-05-07; First posted 2010-05-11 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Castration Resistant Prostate Cancer
Keywords: Castration Resistant; Prostate Cancer; OGX-427
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apatorsen; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OGX-427 and Prednisone (Experimental): OGX-427: Starting within 5 days of randomization, three loading doses at 600 mg IV within the first 10 days of initiating treatment, followed by weekly doses of 1000 mg IV Prednisone: 5 mg BID orally starting within 4 days following randomization and at least 24 hours prior to first loading dose of OGX-427
  Interventions: Drug: OGX-427; Drug: Prednisone
- Prednisone (Active Comparator): Control Arm:
  Prednisone: 5 mg BID orally starting within 4 days following randomization
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: OGX-427 — OGX-427: Starting within 5 days of randomization, three loading doses at 600 mg IV within the first 10 days of initiating treatment, followed by weekly doses of 1000 mg IV
  Other Names: Apatorsen
  Arms: OGX-427 and Prednisone
Drug: Prednisone — Control Arm:
  Prednisone: 5 mg BID orally starting within 4 days following randomization
  Experimental Arm:
  Prednisone: 5 mg BID orally starting within 4 days following randomization and at least 24 hours prior to first loading dose of OGX-427
  Other Names: Rayos; Sterapred

SUMMARY:
This study is being offered to patients who have castrate-resistant (also known as hormone-refractory) prostate cancer. The cancer has metastasized or spread outside the prostate area to other parts of the body or has recurred in the pelvic area after treatment.

The purpose of this clinical research study is to determine whether OGX-427 is able to slow the progression of prostate cancer and symptoms of disease when given with prednisone better than when prednisone is given alone in patients with prostate cancer whose disease has spread outside the prostate area.

Research Hypothesis:

That adding OGX-427 to prednisone treatment will produce a progression free rate of 20%.

DETAILED DESCRIPTION:
Prostate cancer is the most common cancer diagnosed and the second most common cause of cancer death in men in North America.

Patients with metastatic disease have a poor prognosis, and although hormonal therapy in the form of medical or surgical castration can induce significant long-term remissions, development of androgen independent disease is inevitable. The current standard of care for CRPC is mainly palliative in its intent, and there are only limited proven treatment options which include: analgesia, radiation, bisphosphonates and chemotherapy such as mitoxantrone or docetaxel, with only the last treatment being associated with an overall survival benefit.

With the early commencement of androgen deprivation therapy and frequent use of PSA for monitoring disease progression, an increasing population of patients with CRPC is now being identified by a rising PSA rather than by new disease or symptoms. Early intervention with chemotherapy is of unknown benefit in these patients, and thus represents an appropriate group for phase II studies to evaluate novel agents with acceptable toxicity profiles.

Heat shock protein (Hsp) family members, including Hsp27, have attracted attention as new therapeutic targets for cancer. Hsp27 is a small, ATP-independent Hsp which is highly conserved across species. Hsp27 is expressed in prostate cancer and other malignancies. Expression of Hsp27 is induced by cell stress, including cytotoxic chemotherapy, radiation therapy, and hormone therapy. Overexpression of Hsp27 confers a resistant phenotype and is implicated in castration resistant progression of prostate cancer.

OGX 427 is a second generation antisense oligonucleotide (ASO) that inhibits expression of Hsp27. A number of in vitro and in vivo pharmacological studies have demonstrated that OGX 427 (or an Hsp27 ASO) has single-agent activity in reducing Hsp27 mRNA and protein, inhibiting cell proliferation, and inducing apoptosis in several human cancer cell lines. OGX 427 has also demonstrated chemosensitizing activity both in vitro and in vivo in combination with several cytotoxic drugs, including docetaxel. In an ongoing Phase I trial, OGX-427 has been administered as a single agent in doses from 200 to 1000 mg with weekly infusions occurring after a loading dose period of three infusions within the first 10 days of initiating treatment. OGX-427 treatment has been well tolerated, with the majority of the adverse events and laboratory toxicities reported being Grade 1 or Grade 2, although a symptom complex of rigors, pruritus, and erythema during or shortly after infusion of drug has required steroid prophylaxis and/or treatment in some patients at higher doses. No maximum tolerated dose has been identified based on toxicity. OGX 427 administration in combination with docetaxel is ongoing in the above-mentioned Phase 1 study.

Low dose corticosteroids have been shown to have some activity against prostate cancer with a beneficial effect on quality of life (QOL). Since chemotherapy for prostate cancer is palliative, low-dose prednisone has been used both as a single agent and added to chemotherapy regimens.

This Phase 2 study has been designed to evaluate the anti-tumor effects of OGX-427 plus low-dose prednisone versus low-dose prednisone alone in men with CRPC who have not previously received chemotherapy for metastatic or locally recurrent disease.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years on the date of consent.
* ECOG performance status of 0 or 1.
* Histological or cytological diagnosis of adenocarcinoma of the prostate.
* Metastatic disease on chest, abdominal, or pelvic CT and/or bone scan for which no curative therapy exists.
* Progression of prostate cancer. Progression is defined by one or more of the following:

  1. Increasing serum PSA level: two consecutive increases in PSA levels documented over a previous reference value obtained at least one week apart. If the third PSA value is less than the second, an additional fourth test to confirm a rising PSA is acceptable. The last confirmation PSA value must be obtained within the 14 days prior to randomization. A minimum starting value of 2.0 ng/mL is required for study randomization.
  2. Progressive measurable disease: at least a 20% increase in the sum of the diameters of measurable lesions over the smallest sum observed or the appearance of one or more new lesions as assessed by CT scan. Measurable lesions are nodal or visceral soft-tissue lesions with nodal lesions ≥ 15 mm in diameter at the shortest axis and visceral/soft-tissue lesions ≥ 10 mm in longest diameter (See Section 6.4).
  3. Bone Progression: appearance of 2 or more new lesions on bone scan (or other imaging).
* All patients who have not had a surgical orchiectomy must continue treatment with LHRH agonist or antagonist to maintain a castrate level of testosterone.
* Patient must fulfill "Prior Therapy" criteria as follows:

  1. Chemotherapy: No prior chemotherapy for metastatic disease is permissible. (Exception: neoadjuvant/adjuvant chemotherapy if received > 12 months prior to randomization.)
  2. Hormone therapy: prior surgical or medical castration therapy is required. Prior treatment with non-steroidal antiandrogens, abiraterone or other experimental hormone therapy (e.g. MDV3100, YAK-700) is allowed provided a minimum of at least 14 days have passed since completing therapy and randomization in the study.
  3. Experimental therapy: prior non-cytotoxic experimental therapy is permitted provided a minimum of at least 14 days has passed since completing therapy prior to randomization.
  4. Radiation: prior external beam radiation is permitted provided a minimum of at least 28 days have passed since completing radiotherapy at the time of randomization (or following disease progression and prior to receiving therapy at the time of cross-over). Exception for radiotherapy: at least 7 days must have passed since completing single fraction of ≤ 800 cGy.
  5. Corticosteroids: prior corticosteroid therapy is permitted. Within 4 days following randomization, all patients must be taking prednisone 5 mg BID.
* Baseline laboratory values as stated below:

  1. ANC ≥ 1.5 x 109 cells /L, platelet count ≥ .100 x 109 /L, and hemoglobin ≥ 9 g/dL without transfusion.
  2. Creatinine ≤ 1.5 x upper limit of normal (ULN).
  3. Total bilirubin ≤ 1.1 x ULN (unless elevated secondary to conditions such as Gilbert's disease).
  4. SGPT (ALT) and SGOT (AST) ≤ 2.5 x ULN.
  5. Castrate serum testosterone level (< 50 ng/dL-or-< 1.7 nmol/L).
* Recovery from all toxicities of prior therapy to ≤ grade 2 by NCI CTCAE, version 3.0. (Exception: any toxicity that in the view of the Investigator is not a clinically significant safety risk for further therapy administration, including, but not limited to: anemia, fatigue, erectile dysfunction, hot flashes, lymphedema of an extremity, dizziness, cough, and urinary incontinence).
* Must be willing to use effective contraception, if of child bearing potential, throughout study treatment and for 3 months after completion of study treatment.
* Must be willing not to change (add or subtract) bone protecting therapy (bisphosphonates and/or denosumab) during the study unless changed for toxicity.
* Written informed consent must be obtained prior to any protocol-specific procedures being performed.

Exclusion Criteria

* Unable to tolerate a dose of 10 mg of prednisone a day.
* Requiring an amount of opioids to control pain > 30 mg of a morphine-equivalent per day.
* Known coagulopathy or actively receiving warfarin (Coumadin) therapy.
* Documented brain metastases, or carcinomatous meningitis, treated or untreated (Brain imaging for asymptomatic patients is not required).
* Current symptomatic cord compression requiring surgery or radiation therapy (once successfully treated and there has been no progression, patients are eligible for the study).
* Active second malignancy (except adequately treated non-melanomatous skin cancer or other solid tumors curatively treated with no evidence of disease > 3 years).
* History of allergic reactions to therapeutic antisense oligonucleotides.
* Uncontrolled medical conditions such as heart failure, myocardial infarction, uncontrolled hypertension, stroke or treatment of a major active infection within 3 months of randomization, as well as any significant concurrent medical illness that in the opinion of the Investigator would preclude protocol therapy.
* Planned concomitant participation in another clinical trial of an experimental agent, vaccine, or device. Concomitant participation in observational studies is acceptable.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2010-09; Primary Completion 2012-10 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Disease Progression | 12 weeks
  The primary efficacy endpoint is defined as the proportion of patients without disease progression at the 12-week evaluation after treatment with prednisone given with or without OGX-427.

CONTACTS AND LOCATIONS:
Overall Officials: Kim N Chi, MD, Study Chair — BC Cancer Agency - Vancouver Center
Locations (6):
- University of Washington/Seattle Cancer Care Alliance, Seattle, Washington, United States
- Canada (5):
  - BC Cancer Agency - Centre for the Southern Interior, Kelowna, British Columbia
  - BC Cancer Agency - Vancouver Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Background] Scher HI, Halabi S, Tannock I, Morris M, Sternberg CN, Carducci MA, Eisenberger MA, Higano C, Bubley GJ, Dreicer R, Petrylak D, Kantoff P, Basch E, Kelly WK, Figg WD, Small EJ, Beer TM, Wilding G, Martin A, Hussain M; Prostate Cancer Clinical Trials Working Group. Design and end points of clinical trials for patients with progressive prostate cancer and castrate levels of testosterone: recommendations of the Prostate Cancer Clinical Trials Working Group. J Clin Oncol. 2008 Mar 1;26(7):1148-59. doi: 10.1200/JCO.2007.12.4487. PMID 18309951
- [Background] Scher HI, Fizazi K, Saad F, Taplin ME, Sternberg CN, Miller K, de Wit R, Mulders P, Chi KN, Shore ND, Armstrong AJ, Flaig TW, Flechon A, Mainwaring P, Fleming M, Hainsworth JD, Hirmand M, Selby B, Seely L, de Bono JS; AFFIRM Investigators. Increased survival with enzalutamide in prostate cancer after chemotherapy. N Engl J Med. 2012 Sep 27;367(13):1187-97. doi: 10.1056/NEJMoa1207506. Epub 2012 Aug 15. PMID 22894553
- [Background] de Bono JS, Logothetis CJ, Molina A, Fizazi K, North S, Chu L, Chi KN, Jones RJ, Goodman OB Jr, Saad F, Staffurth JN, Mainwaring P, Harland S, Flaig TW, Hutson TE, Cheng T, Patterson H, Hainsworth JD, Ryan CJ, Sternberg CN, Ellard SL, Flechon A, Saleh M, Scholz M, Efstathiou E, Zivi A, Bianchini D, Loriot Y, Chieffo N, Kheoh T, Haqq CM, Scher HI; COU-AA-301 Investigators. Abiraterone and increased survival in metastatic prostate cancer. N Engl J Med. 2011 May 26;364(21):1995-2005. doi: 10.1056/NEJMoa1014618. PMID 21612468
- [Background] Ryan CJ, Smith MR, de Bono JS, Molina A, Logothetis CJ, de Souza P, Fizazi K, Mainwaring P, Piulats JM, Ng S, Carles J, Mulders PF, Basch E, Small EJ, Saad F, Schrijvers D, Van Poppel H, Mukherjee SD, Suttmann H, Gerritsen WR, Flaig TW, George DJ, Yu EY, Efstathiou E, Pantuck A, Winquist E, Higano CS, Taplin ME, Park Y, Kheoh T, Griffin T, Scher HI, Rathkopf DE; COU-AA-302 Investigators. Abiraterone in metastatic prostate cancer without previous chemotherapy. N Engl J Med. 2013 Jan 10;368(2):138-48. doi: 10.1056/NEJMoa1209096. Epub 2012 Dec 10. PMID 23228172
- [Background] Chi KN, Kheoh T, Ryan CJ, Molina A, Bellmunt J, Vogelzang NJ, Rathkopf DE, Fizazi K, Kantoff PW, Li J, Azad AA, Eigl BJ, Heng DY, Joshua AM, de Bono JS, Scher HI. A prognostic index model for predicting overall survival in patients with metastatic castration-resistant prostate cancer treated with abiraterone acetate after docetaxel. Ann Oncol. 2016 Mar;27(3):454-60. doi: 10.1093/annonc/mdv594. Epub 2015 Dec 18. PMID 26685010
- [Background] de Bono JS, Oudard S, Ozguroglu M, Hansen S, Machiels JP, Kocak I, Gravis G, Bodrogi I, Mackenzie MJ, Shen L, Roessner M, Gupta S, Sartor AO; TROPIC Investigators. Prednisone plus cabazitaxel or mitoxantrone for metastatic castration-resistant prostate cancer progressing after docetaxel treatment: a randomised open-label trial. Lancet. 2010 Oct 2;376(9747):1147-54. doi: 10.1016/S0140-6736(10)61389-X. PMID 20888992
- [Background] Smith TJ, Khatcheressian J, Lyman GH, Ozer H, Armitage JO, Balducci L, Bennett CL, Cantor SB, Crawford J, Cross SJ, Demetri G, Desch CE, Pizzo PA, Schiffer CA, Schwartzberg L, Somerfield MR, Somlo G, Wade JC, Wade JL, Winn RJ, Wozniak AJ, Wolff AC. 2006 update of recommendations for the use of white blood cell growth factors: an evidence-based clinical practice guideline. J Clin Oncol. 2006 Jul 1;24(19):3187-205. doi: 10.1200/JCO.2006.06.4451. Epub 2006 May 8. PMID 16682719
- [Background] Bubley GJ, Carducci M, Dahut W, Dawson N, Daliani D, Eisenberger M, Figg WD, Freidlin B, Halabi S, Hudes G, Hussain M, Kaplan R, Myers C, Oh W, Petrylak DP, Reed E, Roth B, Sartor O, Scher H, Simons J, Sinibaldi V, Small EJ, Smith MR, Trump DL, Wilding G, et al. Eligibility and response guidelines for phase II clinical trials in androgen-independent prostate cancer: recommendations from the Prostate-Specific Antigen Working Group. J Clin Oncol. 1999 Nov;17(11):3461-7. doi: 10.1200/JCO.1999.17.11.3461. PMID 10550143